CLINICAL TRIAL: NCT06559540
Title: SWIFT RT: Ultra-Hypofractionated vs. Hypofractionated Radiation for Node-Positive Breast Cancer
Brief Title: Ultra-Hypofractionated vs. Hypofractionated Radiation for Node-Positive Breast Cancer
Acronym: SWIFT RT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202407159
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Node-positive Breast Cancer
Keywords: Breast cancer; Radiation; Hypofractionation; QOL; Cosmesis; Toxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hypofractionated radiation (RT) (Active Comparator): Breast/chest wall and nodal radiation (4256 cGy in 16 fractions over 3-4 weeks).
  Interventions: Radiation: Hypofractionated radiation
- Ultra-hypofractionated breast/chest wall and regional nodal radiation (SWIFT RT) (Experimental): Breast/chest wall and nodal radiation (2600 cGy in 5 fractions over 1-2 weeks).
  Interventions: Radiation: Ultra-hypofractionated breast/chest wall and regional nodal radiation

INTERVENTIONS:
Radiation: Hypofractionated radiation — External beam photon therapy with IMRT or VMAT to the breast/chestwall and regional lymph nodes, including supraclavicular, infraclavicular, axillary, and internal mammary nodes,
  Other Names: RT
  Arms: Hypofractionated radiation (RT)
Radiation: Ultra-hypofractionated breast/chest wall and regional nodal radiation — External beam photon therapy with IMRT or VMAT to the breast/chestwall and regional lymph nodes, including supraclavicular, infraclavicular, axillary, and internal mammary nodes
  Other Names: SWIFT RT
  Arms: Ultra-hypofractionated breast/chest wall and regional nodal radiation (SWIFT RT)

SUMMARY:
In breast cancer patients with nodal involvement, numerous studies have demonstrated that adjuvant radiation therapy reduces the risk of local recurrence, regional recurrence, and distant metastases, in addition to improving survival. The dose and fractionation for adjuvant breast radiation therapy has evolved over time, as novel schedules have been compared to the current standard of care. Hypofractionated radiation therapy (266 cGy per fraction x 15-16 fractions over 3 weeks) has been shown to result in equivalent oncologic outcomes, as well as equivalent acute and late toxicity, when compared to standard fractionation (200 cGy per fraction x 25 fractions over 5 weeks). Subsequently, hypofractionated breast radiation has become the current standard of care.

More recently, ultra-hypofractionated breast radiation (520 cGy per fraction x 5 fractions over 1 week) was shown in a randomized trial to be non-inferior to hypofractionated radiation when treating the breast after lumpectomy. However, the efficacy and toxicity of using ultra-hypofractionated radiation therapy when also treating the regional nodes has not been reported. This is important, as there is greater radiation exposure to several normal tissues, such as the arm/shoulder, brachial plexus, normal lymphatics, heart, and lung, when treating the regional nodes.

In this randomized study, the investigators aim to compare the tolerability and efficacy of ultra-hypofractionated breast/chest wall and regional nodal radiation (SWIFT RT) against hypofractionated radiation (RT). The investigators will evaluate acute and late toxicity, oncologic outcomes (including local recurrence, regional recurrence, distant metastasis, and overall survival), cosmesis, and patient-reported quality of life. The investigators will collect blood samples for correlative studies of biomarkers of fibrosis and cardiac toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive carcinoma of the breast. Metaplastic breast cancer is allowed.
* AJCC 8th Edition Stage: cT1-3 primary tumor. cN1-2 or pN1-2.
* Biopsy-proven involved axillary node(s) (either at baseline and/or at time of surgery).
* Undergone either partial mastectomy (with negative final histologic margins (defined as no tumor on ink, after initial surgery or re-excision)) or mastectomy (with negative histologic margins defined as tumor (either invasive or in situ disease) > 2 mm from the final margin).
* Nodal surgery with either sentinel lymph node biopsy or axillary lymph node dissection. Effort to recover the original biopsy-proven node should be performed at time of surgery.
* Systemic therapy (chemotherapy and/or endocrine therapy) should be administered as per standard of care and recommendation of medical oncology. Neoadjuvant and/or adjuvant systemic therapy is allowed. Concurrent endocrine therapy, anti-HER2 therapy, and immunotherapy during RT is allowed.
* All radiation therapy must be planned to be delivered at BJH or a Siteman satellite location.
* Female.
* Age ≥ 18 years at diagnosis.
* ECOG Zubrod performance status 0 or 1.
* English speaker.
* Able to understand and willing to sign IRB-approved written informed consent document.

Exclusion Criteria:

* Presence of distant metastases.
* Diagnosis of nonepithelial breast malignancies such as sarcoma or lymphoma.
* Diagnosis of bilateral breast cancer.
* AJCC cT4 disease, pT4 disease, or any skin involvement on exam or pathology, including dermal LVSI.
* Presence of palpable or radiographically suspicious supraclavicular, infraclavicular, or internal mammary nodes.
* Prior radiation therapy which would have any overlap with current radiation therapy plan.
* Diagnosis of prior breast cancer or diagnosis of current breast cancer more than one year prior to enrollment.
* Diagnosis of systemic lupus erythematosis, scleroderma, or dermatomyositis.
* Diagnosis of a coexisting medical condition which limits life expectancy to < 2 years.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational treatment. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Time between last breast cancer surgery to RT simulation is greater than 10 weeks, or time between completion of chemotherapy to RT simulation is greater than 8 weeks, whichever is performed last prior to RT.
* Planning to undergo concurrent chemotherapy.
* Pregnancy, which will be excluded prior to simulation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2034-04-30 (Estimated); Study Completion 2034-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are free of serious treatment related late toxicity. | Day 91 through 5 year follow-up (estimated to be 5 years and 1 month)
  Toxicities of concern may include lymphedema, radiation pneumonitis, brachial plexopathy, rib fracture, cardiac disease, and breast/chest wall fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Thomas, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu